CLINICAL TRIAL: NCT01639807
Title: A Prospective, Randomized, Controlled Clinical Trial Comparing Topical Medical Therapy With Selective Laser Trabeculoplasty in South Indian Population
Brief Title: Clinical Evaluation of Efficacy of SLT to Topical Medication in Lowering IOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEH/SLT/012/2011
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Glaucoma
Keywords: Open Angle Glaucoma or Ocular hypertension
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- latanoprost 2-8˚ C (Active Comparator): latanoprost(0.005%)stored at 2-8˚ C
  Interventions: Drug: Latanoprost
- SLT (Experimental): Selective laser Trabeculoplasty
  Interventions: Procedure: SLT

INTERVENTIONS:
Drug: Latanoprost — Latanoprost (0.005%) eye drops, once daily in the evening
  Arms: latanoprost 2-8˚ C
Procedure: SLT — Selective Laser Trabeculoplasty
  Arms: SLT

SUMMARY:
The purpose of this study is to compare Selective laser trabeculoplasty (SLT) and topical medications for initial treatment of open-angle glaucoma /Ocular Hypertension based on intraocular pressure reduction, treatment side effects, quality of life measures and costs in South Indian Population.

DETAILED DESCRIPTION:
Selective laser trabeculoplasty (SLT), a lasering procedure, is equal to or better than using medication for lowering eye pressure,leading to a better quality of life and being less costly.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: POAG, PXF glaucoma, pigmentary glaucoma or mixed mechanism POAG with a narrow angle, (if laser PI > 3 months ago) defined by standard examination criteria Adequate visualization of angle structures (i.e. clear media and cooperative patient) On no glaucoma medications OU > 1 month On no systemic medications known to IOP (steroids) Visual acuity > 6/24 OU Age - more than 35 yrs and less than 72 yrs

Exclusion Criteria:

A cumulative lifetime use of eye drops for glaucoma that exceeded 14 days; Used any eye drops for glaucoma in the 3 weeks before baseline I visit (washout from < 14 days of use will be permitted); CIGTS visual field score that exceeds 16 in either eye; Evidence of ocular disease other than glaucoma that might affect the measurements of IOP, assessment of visual function, visual field testing Proliferative diabetic retinopathy Previous intraocular surgery one or both eyes except laser PI more than 3 months ago and cataract extraction with PC IOL more than 4 months ago.

Undergone ophthalmic laser (other than laser PI > 3 months ago), refractive, conjunctival, or intraocular surgery in either eye; Would likely require cataract surgery within 6 months of randomization Current or expected use of corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular Pressure | 24 months
  To assess the mean and percentage reduction of Intra Ocular Pressure.

SECONDARY OUTCOMES:
Quality of life | 24 months
  To assess the visual function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE V PUTHURAN, M.B.B.S, M.S, Principal Investigator — Aravind Eye Hospital,Madurai.
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114